CLINICAL TRIAL: NCT01318551
Title: Investigation of Pharmacokinetics, Safety, Tolerability, and Pharmacodynamic Effects of BAY85-3934 in Male and Female Subjects With Renal Impairment and in Age- and Weight-matched Healthy Subjects Following a Single Oral Dose of 20 mg and 40 mg (Optional) BAY 85-3934 Administered as Tablets in a Single-center, Non-randomized, Non-controlled, Non-blinded, Observational Study With Group Stratification
Brief Title: Single Dose Group Stratified Study in Renal Impaired and Healthy Aged and Gender Matched Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15557; 2011-000055-16 (EudraCT Number)
Record Dates: First submitted 2011-03-10; First posted 2011-03-18 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Anemia
Keywords: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: BAY85-3934
- Arm 2 (Experimental)
  Interventions: Drug: BAY85-3934
- Arm 3 (Experimental)
  Interventions: Drug: BAY85-3934

INTERVENTIONS:
Drug: BAY85-3934 — single dose, 20 mg
  Arms: Arm 1
Drug: BAY85-3934 — single dose, 40 mg (optional)
  Arms: Arm 2
Drug: BAY85-3934 — single dose, 80 mg (optional)
  Arms: Arm 3

SUMMARY:
Safety, tolerability, pharmacokinetics and pharmacodynamics will be investigated in a single dose group stratified study in renal impaired and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent must be signed before any study-specific tests or procedures are done.
* Female subjects with no child-bearing potential (postmenopausal women with 12 months of spontaneous amenorrhea or with 6 months of spontaneous amenorrhea and serum FSH concentrations >30 mIU/mL, women with 6 weeks post bilateral ovariectomy, woman with bilateral tubal ligation, and women with hysterectomy).
* Male subjects who agree to use 2 forms of effective contraception during the study and for 12 weeks after receiving the study drug. This must include a condom with spermicide gel for 21 days after drug administration.
* Male subjects who agree not to act as sperm donors for 12 weeks after dosing.
* Age: ≥18 and ≤79 years at the pre-study visit.
* Body mass index (BMI): ≥18 and ≤34 kg/m2.
* Ethnicity: white.
* • Subjects participating in this trial and having received 20 mg BAY 85 3934 are encouraged to participate in the following optionally 40 mg and 80 mg study parts.
* Ability to understand and follow study-related instructions.
* For subjects with renal impairment:

  * In diseased subjects: CLCR <90 mL/min determined from a serum creatinine control.
  * In diseased subjects: stable renal disease, ie a serum creatinine value determined at least 3 months before the pre-study visit during routine diagnostics independently of the study should not vary by more than 20% from the serum creatinine value determined at the pre-study visit.
* For healthy subjects:

  * Mean age and body weight in Group 1 or Group 6 or Group 11 (control group, healthy subjects) and Groups 2 to 5 and Groups 7 to 10 and Groups 12 to 15 should not vary by more than +10 years and +10 kg, respectively..
  * In diseased subjects: CLCR ≥90 mL/min determined from a serum creatinine control.

Exclusion Criteria:

* Participation in another clinical trial during the preceding 3 months for multiple-dose studies and 1 month for single-dose studies; (final examination from previous study to first treatment of new study).
* Exclusion periods from other studies or simultaneous participation in other clinical studies.
* Donation of >100 mL of blood within 4 weeks before the first study drug administration or >500 mL in the preceding 3 months.
* Medical disorder that would impair the subject's ability to complete the study in the opinion of the investigator.
* Severe infection or any clinically significant illness within 4 weeks prior to dosing.
* Known hypersensitivity to the study drugs (active substances, or excipients of the preparations).
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies.
* Positive results for hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibodies (HCV Ab), human immune deficiency virus antibodies (HIV 1/2 Ab).
* Regular use of recreational drugs, eg carnitine products, anabolics.
* Regular daily consumption of ≥ 0.5 L of usual beer or the equivalent quantity of approximately 20 g of alcohol in another form.
* Suspicion of drug or alcohol abuse.
* Positive urine drug screening.
* Regular daily consumption of >25 cigarettes.
* Criteria which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the subject's safety.
* Use of medication within the 2 weeks preceding the study which could interfere with the investigational product.
* For subjects with renal impairment:

  * Acute renal failure.
  * Acute nephritis.
  * Nephrotic syndrome.
  * Any organ transplant < 1 year before participation in this study.
  * Failure of any other major organ system other than the kidney.
  * Relevant impairment in liver function of by option of the investigator.
  * Pre-existing diseases for which it can be assumed that the absorption of the study drugs will not be normal (ie relevant malabsorption, chronic diarrhea).
  * Diastolic blood pressure (DBP) >100 mmHg and/or systolic blood pressure (SBP) >180 mmHg (at the pre-study examination; readings taken at the end of the dosing interval of antihypertensive medication, if any).
  * Heart rate <45 or >100 BPM for subject aged 18 to ≤50 years and <55 or >110 BPM for subject aged >50 to ≤79 years at screening visit.
  * Significant uncorrected rhythm or conduction disturbances such as a second- or third-degree AV block without a cardiac pacemaker or episodes of sustained ventricular tachycardia, or by option of the investigator.
  * Diagnosed malignancy within the past 5 years.
  * Psychiatric disorders which may disable the subjects to consent.
  * Change in chronic medications <4 weeks prior to dosing.
  * Concomitant use of any medication except medications necessary for the treatment of the kidney disease or related complications.
* For healthy subjects

  * Subjects with conspicuous findings in medical history or pre-study examination by option of the investigator.
  * A history of relevant diseases of vital organs, of the central nervous system or other organs.
  * Pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal.
  * Systolic blood pressure <100 mmHg or >145 mmHg.
  * Diastolic blood pressure >95 mmHg.
  * Heart rate <45 or >95 BPM for subject aged 18 to ≤50 years and <55 or >95 BPM for subject aged >50 to ≤79 years at screening visit.
  * Clinically relevant findings in the ECG such as a second- or third-degree AV block, clinically relevant prolongation of the QRS complex >120 ms or of the QTc interval >450 ms for men and >470 ms for women of by option of the investigator.
  * Clinically relevant deviations of the screened laboratory parameters in clinical chemistry, hematology, or urinalysis from reference range of by option of the investigator.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-03-16 (Actual); Primary Completion 2013-09-05 (Actual); Study Completion 2014-08-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 4 weeks

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of BAY85-3934 | Day 0 to day 4
Peak Plasma Concentration (Cmax) of BAY85-3934 | Day 0 to day 4
Dose-normalized area under the plasma concentration-time curve (AUCnorm) of BAY85-3934 | Day 0 to day 4
Dose- and body weight-normalised Cmax (Cmax-norm) of BAY85-3934 | Day 0 to day 4

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Kiel, Schleswig-Holstein, Germany

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/